CLINICAL TRIAL: NCT05486039
Title: Adaptation of Mattresses Made With Different Materials to Personal Anthropometry Values and Body Postures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Turkmen, Asst.Prof, Çankırı Karatekin University
Other Study IDs: 28-06-22/26
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Pressure Ulcer; Sleep Disorder; Spine Degeneration; Body Structure, Altered From Its Original Anatomical Structure
MeSH Terms: conditions — Pressure Ulcer; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Normal Posture
  Interventions: Behavioral: Changing behaviour
- Lordotic Posture
  Interventions: Behavioral: Changing behaviour
- Sway Back Posture
  Interventions: Behavioral: Changing behaviour
- Hypolordotic Back Posture
  Interventions: Behavioral: Changing behaviour
- Head Anterior Tilt Posture
  Interventions: Behavioral: Changing behaviour
- Scoliotic Posture
  Interventions: Behavioral: Changing behaviour
- Kyphotic Posture
  Interventions: Behavioral: Changing behaviour

INTERVENTIONS:
Behavioral: Changing behaviour — Changing the lying position and mattress system

SUMMARY:
Sleep disorders affect 40% of the adult population each year and are often associated with morbidity and mortality (Kripke et al., 2002; F.-Z. Low et al., 2017). Sleep quality plays a vital role in the overall quality of our lives. Therefore, a good sleep helps to create a quality life rhythm. A quality sleep reduces fatigue and increases physical regeneration (Khaleghipour et al., 2015). Poor sleep quality is due to various environmental factors such as temperature, light, noise and bed quality (Lei et al., 2009). It has been reported that 7% of sleep problems are caused by inappropriate mattresses that affect the load on the spine during sleep (F. Z. Low et al., 2017). Body contact pressure is a measure of the distribution of body weight across the body surface in contact with the mattress. A well-designed mattress usually has the ability to minimize high pressure points applied to the body. However, if the bed is not suitable for the person, pressure sores may develop in the body parts where pressure is intense (Cullum et al., 2004). The areas most affected by high pressure are usually the hips, shoulders and back, which can affect sleep quality and result in drowsiness or body stiffness throughout the day (Jacobson et al., 2002). A recent study by Bae and Ko compared the bed positions of hospital beds and found that a head-to-foot angle of 30° is the best position to reduce the likelihood of decubitus ulcers occurring in patients in high-pressure risk areas (Bae & Ko, 2013). In the light of previous studies, it has been observed that there is no study comparing many bed types designed using different materials for individual-specific postures. Biomechanical comparison of these bedding materials in individuals with different posture types and sleeping in different sleeping positions will allow us to provide new insights into their pressure distribution abilities. The aim of this study is to measure the effect of mattresses made of different mattress materials on body contact pressure profiles in individuals with different postures in various sleeping positions. It will be evaluated using maximum body pressure and pressure distribution as outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in research

Exclusion Criteria:

* Having a history of back, shoulder or neck pain in the last 6 weeks
* Having a surgical operation in the last 8 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 210 participants (105 women, 105 men) between the ages of 18-85 with 7 different posture types (Normal posture, Lordotic posture, "sway back" posture, straight waist posture, head forward posture, scoliotic posture and kyphotic posture) will be included in this study. .
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of Total Body Pressure | 40 minutes
  A pressure mat sensor (Pressure Mapping Sensor 5400N, Tekscan, Boston, MA) will first be calibrated on different beds using constant weights and then used to capture body contact pressure profiles in a video format for 6 minutes per stop at a sampling rate. 4 Hz Collected data will be edited in Matlab (MathWorks, Natick, MA) format for later recording. The posture screen analysis system will be used to determine the posture type of individuals.

SECONDARY OUTCOMES:
Pittsburg Health Quality Index | 40 minutes
  The Pittsburg Sleep Quality Scale will be used to obtain more detailed data on current sleep quality from individuals (Buysse et al., 1989).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Cullum N, McInnes E, Bell-Syer SE, Legood R. Support surfaces for pressure ulcer prevention. Cochrane Database Syst Rev. 2004;(3):CD001735. doi: 10.1002/14651858.CD001735.pub2. PMID 15266452
- [Result] Jacobson BH, Gemmell HA, Hayes BM, Altena TS. Effectiveness of a selected bedding system on quality of sleep, low back pain, shoulder pain, and spine stiffness. J Manipulative Physiol Ther. 2002 Feb;25(2):88-92. doi: 10.1067/mmt.2002.121410. PMID 11896375
- [Result] Kripke DF, Garfinkel L, Wingard DL, Klauber MR, Marler MR. Mortality associated with sleep duration and insomnia. Arch Gen Psychiatry. 2002 Feb;59(2):131-6. doi: 10.1001/archpsyc.59.2.131. PMID 11825133
- [Result] Low FZ, Chua MC, Lim PY, Yeow CH. Effects of Mattress Material on Body Pressure Profiles in Different Sleeping Postures. J Chiropr Med. 2017 Mar;16(1):1-9. doi: 10.1016/j.jcm.2016.09.002. Epub 2016 Oct 21. PMID 28228692